CLINICAL TRIAL: NCT05677477
Title: The Effect of Hybrid Simulation on Nursing Students' Ability to Evaluate Neonatal Physiological Jaundice: A Randomized Controlled Trial
Brief Title: The Effect of Hybrid Simulation on Evaluating Neonatal Jaundice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Aylin PEKYİGİT, Research Assistant, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CKU
Record Dates: First submitted 2022-12-05; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Nursing Education
Keywords: Nursing education; hyperbillirubinemia; simulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/Treatment (Experimental): In the implementation process of the research, knowledge tests will be applied as pre-test and post-test, and training will be given to the mother who has a baby with physiological jaundice. In the study, the scenario of the mother with a baby with jaundice will be implemented only with the intervention group
  Interventions: Other: simulation training
- Control (No Intervention): During the application process of the research, knowledge tests will be applied as pre-test and post-test.

INTERVENTIONS:
Other: simulation training — A mother scenario with a baby with physiological jaundice will be implemented with the intervention group.
  Arms: Intervention/Treatment

SUMMARY:
This study will be conducted as a single-blind randomized control group intervention trial to determine the effectiveness of the hybrid simulation method using standard patient and low-fidelity baby simulators in the intervention of nursing students for neonatal physiologic jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the course
* Had not taken this course before
* Accepted to participate in the research

Exclusion Criteria:

* Have any records of absence
* Taken this course before
* Graduate of health vocational high school

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Student Information Form and First Knowledge Test | One week before Simulation (First week)
  Student Information Form (First Knowledge Test-Before Simulation): In this form, which was created by the researcher by scanning the literature, did he choose the student's number, age, gender, graduated high school, nursing department willingly, did he get information about the simulation before, did he get information about neonatal jaundice? ? The questions are included. In the same survey, there is the "Newborn Physiological Jaundice Assessment Test" consisting of 25 questions created by the researchers. In this questionnaire, there are statements regarding the physiological jaundice of the newborn. Students were asked to mark one of the options "Yes", "No" or "I don't know" for these statements. This form was applied to the students as a pre-test. After the pretest, the subject was explained about the physiological jaundice of the newborn.
  This form was filled by both the experimental and control groups.
Jaundice case checklist form | During simulation (Second week)
  Jaundice case checklist form (During simulation): This checklist was created by the researcher. There are statements for learning objectives set to evaluate neonatal jaundice. These expressions are "did", "did not" and "partially did". The behavior of the student during the simulation was evaluated by the researcher and his peers. After the simulation, the student was asked to evaluate himself on this form and fill out the form.
Second Student Knowledge Test | Two weeks after simulation (Fourth week)
  Second Student Knowledge Test (After the Simulation): 2 weeks after the simulation application, the "Newborn Physiological Jaundice Assessment Test" was applied to both the control and experimental groups. In addition to this test, "Student Satisfaction and Self-Confidence Scale in Learning" and "Simulation Design Scale" were applied to the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Müjgan Onarıcı, Study Chair — Çankırı Karatekin University; Tuğba Yıldırım, Study Chair — Çankırı Karatekin University
Locations (1):
- Çankırı Karatekin Üniversitesi, Çankiri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Choi YJ. Exploring experiences of psychiatric nursing simulations using standardized patients for undergraduate students. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Sep;6(3):91-5. doi: 10.1016/j.anr.2012.07.001. Epub 2012 Jul 20. PMID 25030974